CLINICAL TRIAL: NCT05959538
Title: Building Regulation in Dual Generations (BRIDGE) 2022-2025
Brief Title: Building Regulation in Dual Generations 2022-2025
Acronym: BRIDGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRIDGE 2022-2025
Record Dates: First submitted 2023-06-08; First posted 2023-07-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2023-05

CONDITIONS: Maternal Depression; Self-Regulation, Emotion; Child Mental Disorder; Child Development
Keywords: maternal depression; childhood development; child psychopathology; emotion regulation; parenting; stress; prevention science
MeSH Terms: conditions — Emotional Regulation; Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: The study will recruit a group of caregivers in which the caregiver meets the current criteria for elevated symptoms of psychological distress as measured by a score of 9 and above on the Patient Health Questionnaire 9-item. Eligible female caregivers (mothers, grandmothers, aunts, guardians) will be randomly assigned to one of three intervention arms, which will occur concurrently over 16-weeks. One arm will incorporate intervention materials from Dialectical Behavior Therapy (DBT) and parent skills training (BRIDGE), another will provide DBT only, while the third will provide community family support services as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Building Regulation in Dual Generations (BRIDGE; DBT + Parenting) (Experimental): The BRIDGE program is a manualized therapy that provides participants with parenting and DBT skills through video training modules and in-group sessions. Participants in the BRIDGE arm will participate in 16 weeks of 20-30 minute DBT and parenting skills training that will be delivered asynchronously via video (participants will access these by logging onto a password protected website). The BRIDGE condition also includes weekly synchronous 1-hour virtual group therapy sessions as well as DBT and parenting skills worksheets to complete between sessions.
  Interventions: Behavioral: Building Regulation in Dual Generations (BRIDGE)
- Dialectical Behavioural Skills Training (DBT) (Active Comparator): Participants in the DBT arm will participate in 16 weeks of DBT skills training through weekly, synchronous 1.5-hour virtual group therapy sessions. Participants will also be asked to complete worksheets on the content between sessions.
  Interventions: Behavioral: Dialectical Behavioural Therapy Skill Training
- Services-As-Usual (SAU) (No Intervention): Participants in the SAU arm will receive a list of local mental health and parenting resources, curated by our research team. Participants can access any intervention or resource participants would like throughout the duration of the program.

INTERVENTIONS:
Behavioral: Building Regulation in Dual Generations (BRIDGE) — The BRIDGE intervention includes 16 weeks of 20-30 minute DBT and parenting skills training videos, delivered asynchronously via an online website requiring a participant login. Video content was drawn from concepts outlined in the DBT Skills Training Manual 2nd Edition (Linehan, 2015). Parenting videos will provide mothers with parenting skills education based on best practices in evidence-based positive parenting interventions (e.g., Parent Management Training, Positive Parenting, Kazdin, 1997; Sanders et al., 2014). The BRIDGE condition also includes weekly synchronous 1-hour virtual group therapy sessions and worksheets to complete weekly (as an opportunity to practice skill use). The clinical team will consist of two Master's or PhD level clinical psychology trainees and a parent peer coach. Mood tracking will be completed using a brief weekly survey, including questions on depression, parenting stress, positive mood, and recent stressful experiences.
  Arms: Building Regulation in Dual Generations (BRIDGE; DBT + Parenting)
Behavioral: Dialectical Behavioural Therapy Skill Training — Participants in the DBT arm will participate in 16 weeks of DBT skills training only led by two Master's or PhD level clinical psychology trainees. Participants in the DBT Skills condition will participate in a skills group which follows the DBT Skills Training Manual 2nd Edition (Linehan, 2015) through weekly, synchronous 1.5-hour virtual group therapy sessions. Mindfulness, Emotion Regulation, Distress Tolerance, and Interpersonal Effectiveness skill domains will be covered. Participants will be asked to complete worksheets between sessions to practice using skills, and will be asked to complete a Diary Card to track DBT skills use each week (Linehan, 2015). Mood tracking will be completed using a brief weekly survey including questions on depression, parenting stress, positive mood, and recent stressful experiences.
  Arms: Dialectical Behavioural Skills Training (DBT)

SUMMARY:
This randomized control trial aims to investigate whether a novel intervention, the "Building Regulation in Dual Generations (BRIDGE)" program, improves mental wellness and parenting practices among mothers of 3 to 5-year-old children who have elevated symptoms of depression. The main two questions this study aims to answer are:

* Does participation in the BRIDGE program reduce maternal depression symptoms?
* Does participation in the BRIDGE program improve children's mental health?

Researchers will compare the BRIDGE intervention to an established mental health intervention (i.e., Dialectical Behaviour Therapy skills group) and to a services-as-usual control group to see if participation in BRIDGE leads to greater improvements than either the general mental health treatment or community services as usual.

Participants will:

* Complete a set of questionnaires pre- and post-intervention, and at 6-month follow-up.
* Complete a virtual assessment with their child at pre- and post-intervention.
* Be randomized to BRIDGE, Dialectical Behavioural Therapy(DBT) skills group, or a services-as-usual control group.
* Participate in the 16-week BRIDGE or DBT Skills only group, if randomized to either of these groups. If they are randomized to services-as-usual they will receive a list of community resources they can access.
* Complete weekly symptom monitoring via questionnaires, if randomized to BRIDGE or DBT Skills
* Wear a Fitbit device during pre- and post-intervention, as well as throughout the 16-week intervention period.

DETAILED DESCRIPTION:
Diagnosed in 10-15% of children worldwide, childhood mental illness [MI] remains a prominent public health concern. Early exposure to maternal depression is a notable risk factor for the development of childhood MI. Maternal depression is most common in the first few years following childbirth, and clinically significant depressive symptoms are on the rise, with recent estimates at 26.9% for mothers worldwide. This increase highlights the current and critical need for interventions to address maternal depression and the prevention of childhood MI concurrently.

To simultaneously address maternal and child MI, the Building Regulation in Dual Generations (BRIDGE) group-based intervention was created. BRIDGE aims to increase intergenerational emotion regulation by pairing Dialectical Behaviour Therapy (DBT) skills training with a theoretically aligned parenting skills program. DBT has been shown to be a propitious transdiagnostic treatment for underlying mechanisms of psychopathology, including emotion regulation difficulties common in depression, anxiety, and traumatic stress.

Developmentally supportive parenting requires mothers to have the ability to regulate emotions effectively; in so doing, a mother can simultaneously limit over-reactive responses within themselves and towards their child, as well as teach their child about emotions. These objectives map nicely to the skills being learned in DBT. Within BRIDGE, the aligned parenting content also includes best-practice behaviour management training techniques, such as creating positive family routines and using positive reinforcement, framed within the context of DBT skills. The integration of DBT with parenting programs in BRIDGE is a promising approach for addressing intergenerational needs.

The current study will expand on previous evaluations of BRIDGE by conducting a randomized controlled trial (RCT) comparing (1) BRIDGE (DBT skills training + Parenting Skills), (2) DBT (DBT skills training only), and (3) services as usual (SAU). Our primary aim is to examine the effects of BRIDGE on maternal depression and child MI symptoms. We hypothesize that participants who receive the BRIDGE and DBT interventions will report fewer depressive symptoms than participants in the SAU group. Participants who receive the BRIDGE intervention are hypothesized to report fewer child MI symptoms than those in the DBT and SAU groups.

A secondary aim of this study is to evaluate the efficacy of BRIDGE in reducing parenting stress and harsh parenting. Participants who receive the BRIDGE intervention are hypothesized to show lower levels of parenting stress and harsh parenting than those in the DBT and SAU groups.

Interim analyses of primary and secondary outcomes will be conducted at the mid-way point of the RCT, when approximately 90 participants have completed the post-intervention questionnaires (T2). Minor changes in intervention delivery (e.g., offering optional in-person group therapy, updating DBT homework, changing video production) may be made based on results from interim analyses. Any changes to intervention delivery will be documented in a protocol deviation document.

Additional aims of the RCT are to examine the effects of BRIDGE and DBT on family relationships, other service use (e.g., hospital visits, interactions with police), and maternal psychopathology symptoms. The investigators hypothesize that mothers who receive the BRIDGE or DBT intervention will report lower psychopathology symptoms, reduced service use, and improved family relationship quality. The investigators will also assess participants' engagement in each intervention.

Exploratory outcomes of observed maternal sensitivity and child emotion regulation will also be examined via remote Zoom assessments. The investigators hypothesize that mothers in the BRIDGE group will show greater maternal sensitivity and that their children will demonstrate improved emotion regulation, more than those in the DBT or SAU groups.

Additional exploratory outcomes will come from physiological feedback and coparent participation. Physiological indices of wellbeing (e.g., sleep and daily activity) will be measured via Fitbits that mothers will wear during the program. The investigators hypothesize that participants who receive the BRIDGE or DBT interventions will display improved sleep quality and reduced sedentary behaviour.

The investigators will invite participants' co-parents to complete questionnaires on their own mental health and family relationships. Inviting co-parents to complete questionnaires during this trial is exploratory and will allow us to evaluate the feasibility of including assessments of co-parents in future trials. The investigators hypothesize that some spill-over effects of the BRIDGE and DBT interventions may occur, such that co-parents of participants in either intervention group will show fewer MI symptoms and improved family relationship quality.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one 3-5-year-old child.
* Residing in Manitoba or British Columbia, Canada.
* Report elevated symptoms of depression (PHQ-9 score ≥10) at the eligibility screener, pre-randomization.
* Self-identify as being comfortable understanding, speaking and reading English.
* Self-identify as having internet access.
* Report being available to attend telehealth groups.
* Report being willing to complete pre- and post-intervention questionnaires.

Exclusion Criteria:

* Mothers who report a suicide attempt in the past year or who have engaged in self-harm that required medical attention in the past 6 months will not be eligible to participate in the study, as the BRIDGE program is not intended to address these mental health needs.
* In addition, mothers who report a diagnosis of, or treatment for, Post-Traumatic Stress Disorder, Alcohol Use Disorder, Substance Use Disorder, or Psychotic Disorder in the last year will be followed up with a senior clinician to evaluate whether the BRIDGE program would be suitable for their needs. If the clinician (through consultation with clinical leads) indicates that the participant will be able to participate and engage in BRIDGE and/or DBT as the program is to be delivered, they will be considered eligible. Some participants may be encouraged to follow-up with group clinicians to ensure their mental health needs are being managed appropriately within or outside of the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The terms "mother" and "maternal" will be used throughout this paper to describe all participants; however, anyone who self-identifies as a mother or female primary caregiver (e.g., grandmothers raising grandchildren, gender diverse caregivers who identify as mothers) will be eligible to participate.
Enrollment: 197 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Change in depression symptoms | The PHQ-9 will be assessed during eligibility screening, pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Depressive symptoms will be measured using the PHQ-9. The PHQ-9 is a 9-item self-report questionnaire with possible scores ranging from 0 to 27, with higher scores indicating greater symptom severity.
Change in child mental illness symptoms | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Changes in child mental illness symptoms will be assessed using the Child Behaviour Checklist (CBCL). The CBCL is a parent-report questionnaire that measures child functioning across internalizing and externalizing symptoms. The CBCL contains 113 items, with scores ranging from 0-226. Higher scores indicated greater symptom severity.

SECONDARY OUTCOMES:
Change in Parenting stress | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Parenting stress will be measured using the Parenting Stress Index-Short Form (PSI-SF). The PSI-SF is a self-report questionnaire that requires respondents to answer questions regarding their overall experience with parenting stress using a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Scores range from 36-180. Higher scores indicate higher levels of stress.
Change in harsh parenting | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Harsh parenting will be measured using the Overreactivity subscale of the Parenting Scale (PS). The Overreactivity subscale contains 10 items related to harsh parenting behaviours. Harsh parenting includes expressing inappropriate anger, irritability, or meanness towards one's child. Totals scores range from 10 to 70, with higher scores indicating higher levels of harsh parenting.

OTHER OUTCOMES:
Change in couples' relationship satisfaction. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Using the Couples Satisfaction Index (CSI-4), the investigators will examine participants' satisfaction with their romantic relationships. The CSI-4 contains 4 -items. Total scores range from 0-21, with higher scores indicating greater relationship satisfaction.
Change in social support. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  The Multidimensional Scale of Perceived Social Support (MSPSS) will be used to measure participant's levels of social support from significant others, family, and friends. Scores can range from 12-84. Higher scores indicated higher levels of perceived social support.
Change in parenting practices related to children's negative emotions. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  The Coping with Children's Negative Emotions Scale (CCNES) presents hypothetical scenarios in which a child gets upset or angry. Parents are asked to indicate the degree to which the parent responds to each scenario in 6 theoretically meaningful ways of coping with children's negative emotions. The CCNES has 6 subscales: Problem-Focused Reactions (PRF), Emotion-Focused Reactions (EFR), Expressive Encouragement (EE), Minimization Reactions (MR), Punitive Reactions PR), and Distress Reactions (DR). Each subscale has a score range from 12-84. Higher scores on each subscale represent higher levels of that type of parenting response (e.g., high expressive encouragement scores represent parenting practices in which parents encourage their children to express their emotions).
Change in anxiety symptoms. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Anxiety symptoms will be measured using the Generalized Anxiety Disorder 7-Item Scale (GAD-7). The GAD-7 contains 7 items with possible scores ranging from 0 to 21. Higher scores represent higher levels of anxiety symptoms.
Change in self-compassion. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  The Self-Compassion Scale-Short Form (SCS-SF) will be used to measure changes in participants' self-compassion. Possible scores range from 12-60, with higher scores indicating high levels of self-compassion.
Change in anger. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Changes in anger will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Anger subscale. The subscale contains 5-items with scores ranging from 5-25. Higher scores indicate more anger.
Change in sleep disturbance. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  The Patient-Reported Outcomes Measurement Information System-Sleep Disturbance Subscale Short Form will be used to measure change in sleep disturbances. The subscale contains 8 items. Total scores range from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
Change in alcohol use. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  The Alcohol Use Disorder Identification Test (AUDIT) will be used to measure participants' use of alcohol. The AUDIT contains 10 question and scores may range from 10 to 40. Higher scores indicate greater hazardous or harmful alcohol consumption.
Change in cannabis use. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  The Cannabis Use Disorder Identification Test (CUDIT) will be used to measure participants' cannabis use. The scale contains 8 items. Scores may range from 0 to 32. Higher scores indicate more hazardous cannabis use.
Change in observed maternal sensitivity | Assessed at pre-intervention (T1) and within a month following the intervention.
  Participants and their children will attend pre- and post-intervention virtual assessments, where they will be asked to complete a free-play and clean-up task, which will be video recorded. Video recordings of the task will be coded using the Maternal Q-Sort developed by Pederson et al. (1999).
Change in observed child emotional regulation | Assessed at pre-intervention (T1) and within a month following the intervention.
  Participants and their children will attend pre- and post-intervention virtual assessments, where children will be asked to complete an emotion-inducing task, which will be video recorded. Video recordings of the task will be coded using a coding scheme developed by the research team.
Change in health and social services use. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  A self-report scale created for use in this project will assess participants' use of 14 types of health and social services in the previous 3 months. The scale does not produce a total score; rather, the scale asks participants if they had accessed services, and if yes, the frequency of their use of those services.
Change in recent stressful experiences. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  The Recent Stressful Experiences checklist (RSE) was developed by study authors, based on recommendations from the JBP Research Network on Toxic Stress at the Harvard's Center on the Developing Child, to measure familial exposure to various stressors which may affect participants (2022). The scale contains two items which ask about various stressors that participants may have experienced. Each of these items' scores can range from 0 to 10, with higher scores indicating more stressful experiences. The scale also contains five items assessing participants' ability to cope with stressful events. Scores for these five questions range from 4-21, with higher scores indicating a greater ability to cope with stress.
Program engagement | Measured weekly throughout the 16-week program and immediately after the intervention (T2).
  Program engagement will be assessed in a variety of ways. In both the BRIDGE and DBT Skills-only groups, clinicians will take attendance during therapy sessions. In the BRIDGE group, the investigators will extract aggregate data on the number of views on the psychoeducational videos using Google Analytics. At post-intervention, the investigators will ask participants to report about their use of the videos, homework assignments, and mood tracking throughout the intervention. Participants in the BRIDGE group will also complete a program acceptability questionnaire at post-intervention which was created by the investigators for this project. The program acceptability questionnaire asks participants to rate how important various program components were to them and includes several open-ended questions for participants to describe their experiences in the program.
Change in physical activity | Measured at pre-intervention (T1), throughout the 16-week intervention, and for a month following the intervention.
  Physical activity will be assessed via step-count using Fitbit devices worn by participants.
Change in sleep quality | Measured at pre-intervention (T1), throughout the 16-week intervention, and for a month following the intervention.
  Sleep quality will be measured throughout the intervention using Fitbit devices worn by participants.
Change in sleep duration | Measured at pre-intervention (T1), throughout the 16-week intervention, and for a month following the intervention.
  Sleep duration will be measured throughout the intervention using Fitbit devices worn by participants.
Change in heart rate | Measured at pre-intervention (T1), throughout the 16-week intervention, and for a month following the intervention.
  Heart rate will be measured throughout the intervention using Fitbit devices worn by participants.
Change in co-parents' depression symptoms. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Co-parents of participants will be invited to complete a set of questionnaires. The PHQ-9 will be used to measure co-parents' depression symptoms. The PHQ-9 is a 9-item self-report questionnaire with possible scores ranging from 0 to 27, with higher scores indicating greater symptom severity.
Change in co-parents' rating of child behaviour. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Co-parents of participants will be invited to complete a set of questionnaires. The CBCL will be used to assess co-parents' ratings of child behaviour. The CBCL is a parent-report questionnaire that measures child functioning across internalizing and externalizing symptoms. The CBCL contains 113 items, with scores ranging from 0-226. Higher scores indicated greater symptom severity.
Change in co-parents' parenting stress. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Co-parents of participants will be invited to complete a set of questionnaires. The PSI-SF will be used to assess co-parents' parenting stress. The PSI-SF is a self-report questionnaire that requires respondents to answer questions regarding their overall experience with parenting stress using a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Scores range from 36-180. Higher scores indicate higher levels of stress.
Change in co-parents' harsh parenting. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Co-parents of participants will be invited to complete a set of questionnaires PS Overreactivity. Harsh parenting will be measured using the Overreactivity subscale of the Parenting Scale (PS). The Overreactivity subscale contains ten items related to harsh parenting behaviours. Harsh parenting includes expressing inappropriate anger, irritability, or meanness towards one's child. Total scores range from 10 to 70, with higher scores indicating higher levels of harsh parenting.
Change in co-parents' couples' satisfaction. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Co-parents of participants will be invited to complete a set of questionnaires. Using the Couples Satisfaction Index (CSI-4) the investigators will examine co-parents' satisfaction with their romantic relationships. The CSI-4 contains 4 -items. Total scores range from 0-21, with higher scores indicating greater relationship satisfaction.
Change in co-parents' social support. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Co-parents of participants will be invited to complete a set of questionnaires. The MSPSS will be used to measure co-parents' social support. Scores can range from 12-84. Higher scores indicated higher levels of perceived social support.
Change in co-parents' parenting practices related to children's negative emotions. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Co-parents of participants will be invited to complete a set of questionnaires. The Coping with Children's Negative Emotions Scale (CCNES) presents hypothetical scenarios in which a child gets upset or angry. Parents are asked to indicate the degree to which the parent responds to each scenario in 6 theoretically meaningful ways of coping with children's negative emotions. The CCNES has 6 subscales: Problem-Focused Reactions (PRF), Emotion-Focused Reactions (EFR), Expressive Encouragement (EE), Minimization Reactions (MR), Punitive Reactions PR), and Distress Reactions (DR). Each subscale has a score range from 12-84. Higher scores on each subscale represent higher levels of that type of parenting response (e.g., high expressive encouragement scores represent parenting practices in which parents encourage their children to express their emotions).
Change in co-parents's self-compassion. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Co-parents of participants will be invited to complete a set of questionnaires. The SCS-SF will measure co-parents' self-compassion. Possible scores range from 12-60, with higher scores indicating high levels of self-compassion.
Change in co-parents' anxiety symptoms. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Co-parents of participants will be invited to complete a set of questionnaires. Anxiety symptoms will be measured using the GAD-7. The GAD-7 contains 7 items with possible scores ranging from 0 to 21. Higher scores represent higher levels of anxiety symptoms.
Change in co-parents' anger. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Co-parents of participants will be invited to complete a set of questionnaires. Changes in anger will be measured using PROMIS Anger subscale. The subscale contains 5-items with scores ranging from 5-25. Higher scores indicate more anger.
Change in co-parents' sleep disturbances. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Co-parents of participants will be invited to complete a set of questionnaires. The PROMIS-Sleep Disturbance Subscale Short Form will be used to measure change in sleep disturbances. The subscale contains 8 items. Total scores range from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
Change in co-parents' alcohol use. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Co-parents of participants will be invited to complete a set of questionnaires. The Alcohol Use Disorder Identification Test (AUDIT) will be used to measure coparents' use of alcohol. The AUDIT contains 10 question and scores may range from 10 to 40. Higher scores indicate greater hazardous or harmful alcohol consumption.
Change in co-parents' cannabis use. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Co-parents of participants will be invited to complete a set of questionnaires. The Cannabis Use Disorder Identification Test (CUDIT) will be used to measure coparents' cannabis use. The scale contains 8 items. Scores may range from 0 to 32. Higher scores indicate more hazardous cannabis use.
Change in co-parents' recent stressful experiences. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  Co-parents of participants will be invited to complete a set of questionnaires. The Recent Stressful Experiences checklist (RSE) was developed by study authors, based on recommendations from the JBP Research Network on Toxic Stress at the Harvard's Center on the Developing Child, to measure familial exposure to various stressors which may affect participants (2022). The scale contains two items which ask about various stressors that participants may have experienced. Each of these items' scores can range from 0 to 10, with higher scores indicating more stressful experiences. The scale also contains five items assessing participants' ability to cope with stressful events. Scores for these five questions range from 4-21, with higher scores indicating a greater ability to cope with stress.
Change in co-parents' health and social services use. | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3).
  A self-report scale created for use in this project will assess coparents' use of 14 types of health and social services in the previous 3 months. The scale does not produce a total score; rather, the scale asks participants if they had accessed services, and if yes, the frequency of their use of those services.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie R. Roos, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba - Department of Psychology, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
Summary statistics (e.g. questionnaire subscales, socio-demographics, aggregated forum usage data) paired with non-identifiable participant IDs may be shared on data repositories such as the Open Science Framework.
Supporting Information: Study Protocol
Time Frame: Data may become available upon publication of study results, in approximately October 2024.
Access Criteria: Access will be based on the academic journal's level of access and requirements (e.g., subscription). Open access will be preferred at the time of journal selection, as possible, and preprint articles will be submitted online (e.g., psyarxiv.com) as possible based on journal requirements.

REFERENCES:
- [Background] Polanczyk GV, Salum GA, Sugaya LS, Caye A, Rohde LA. Annual research review: A meta-analysis of the worldwide prevalence of mental disorders in children and adolescents. J Child Psychol Psychiatry. 2015 Mar;56(3):345-65. doi: 10.1111/jcpp.12381. Epub 2015 Feb 3. PMID 25649325
- [Background] Shonkoff JP, Fisher PA. Rethinking evidence-based practice and two-generation programs to create the future of early childhood policy. Dev Psychopathol. 2013 Nov;25(4 Pt 2):1635-53. doi: 10.1017/S0954579413000813. PMID 24342860
- [Background] Horwitz SM, Briggs-Gowan MJ, Storfer-Isser A, Carter AS. Persistence of Maternal Depressive Symptoms throughout the Early Years of Childhood. J Womens Health (Larchmt). 2009 May;18(5):637-45. doi: 10.1089/jwh.2008.1229. PMID 19445615
- [Background] Swales DA, Snyder HR, Hankin BL, Sandman CA, Glynn LM, Davis EP. Maternal Depressive Symptoms Predict General Liability in Child Psychopathology. J Clin Child Adolesc Psychol. 2022 Jan-Feb;51(1):85-96. doi: 10.1080/15374416.2020.1723598. Epub 2020 Mar 27. PMID 32216604
- [Background] Wang L, Wu T, Anderson JL, Florence JE. Prevalence and risk factors of maternal depression during the first three years of child rearing. J Womens Health (Larchmt). 2011 May;20(5):711-8. doi: 10.1089/jwh.2010.2232. Epub 2011 Mar 22. PMID 21426237
- [Background] Racine N, Eirich R, Cooke J, Zhu J, Pador P, Dunnewold N, Madigan S. When the Bough Breaks: A systematic review and meta-analysis of mental health symptoms in mothers of young children during the COVID-19 pandemic. Infant Ment Health J. 2022 Jan;43(1):36-54. doi: 10.1002/imhj.21959. Epub 2021 Dec 28. PMID 34962649
- [Background] Delaquis CP, Joyce KM, Zalewski M, Katz LY, Sulymka J, Agostinho T, Roos LE. Dialectical behaviour therapy skills training groups for common mental health disorders: A systematic review and meta-analysis. J Affect Disord. 2022 Mar 1;300:305-313. doi: 10.1016/j.jad.2021.12.062. Epub 2021 Dec 26. No abstract available. PMID 34965396
- [Background] Harley R, Sprich S, Safren S, Jacobo M, Fava M. Adaptation of dialectical behavior therapy skills training group for treatment-resistant depression. J Nerv Ment Dis. 2008 Feb;196(2):136-43. doi: 10.1097/NMD.0b013e318162aa3f. PMID 18277222
- [Background] Zalewski, M., Maliken, A. C., Lengua, L. J., Martin, C. G., Roos, L. E., & Everett, Y. (2020). Integrating dialectical behavior therapy with child and parent training interventions: A narrative and theoretical review. Clinical Psychology: Science and Practice.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kristensen S, Henriksen TB, Bilenberg N. The Child Behavior Checklist for Ages 1.5-5 (CBCL/1(1/2)-5): assessment and analysis of parent- and caregiver-reported problems in a population-based sample of Danish preschool children. Nord J Psychiatry. 2010 May 4;64(3):203-9. doi: 10.3109/08039480903456595. PMID 20085433
- [Background] Abidin, R. R. (1995). Parenting Stress Index (3rd ed.). Odessa, FL: Psychological Assessment Resources.
- [Background] Arnold, D. S., O'leary, S. G., Wolff, L. S., & Acker, M. M. (1993). The Parenting Scale: a measure of dysfunctional parenting in discipline situations. Psychological assessment, 5(2), 137.
- [Background] Funk JL, Rogge RD. Testing the ruler with item response theory: increasing precision of measurement for relationship satisfaction with the Couples Satisfaction Index. J Fam Psychol. 2007 Dec;21(4):572-83. doi: 10.1037/0893-3200.21.4.572. PMID 18179329
- [Background] Fabes, R. A., Eisenberg, N., & Bernzweig, J. (1990). Coping with Children's Negative Emotions Scale (CCNES): Description and scoring. Tempe, AZ: Arizona State University.
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID 22250775
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Adamson SJ, Kay-Lambkin FJ, Baker AL, Lewin TJ, Thornton L, Kelly BJ, Sellman JD. An improved brief measure of cannabis misuse: the Cannabis Use Disorders Identification Test-Revised (CUDIT-R). Drug Alcohol Depend. 2010 Jul 1;110(1-2):137-43. doi: 10.1016/j.drugalcdep.2010.02.017. Epub 2010 Mar 26. PMID 20347232
- [Background] Pederson, D. R., Moran, G., & Bento, S. (1999). Maternal behaviour Q-sort.
- [Derived] Penner-Goeke L, Belows M, Kristjanson A, Andrade BF, Cameron EE, Giuliano R, Katz LY, Kelly LE, Letourneau N, Mota N, Reynolds K, Zalewski M, Pharazyn A, Roos LE. Protocol for a randomized control trial of the Building Regulation in Dual Generations Program (BRIDGE): preventing the intergenerational transmission of mental illness in at-risk preschool children. Trials. 2023 Sep 19;24(1):597. doi: 10.1186/s13063-023-07591-8. PMID 37726821